CLINICAL TRIAL: NCT02145156
Title: Educational Intervention to Minimize Disparities in HPV Vaccination
Brief Title: Educational Intervention to Minimize Disparities in Humanpapillomavirus Vaccination
Acronym: HPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 14-0402; PCORI 1455 (Other Grant/Funding Number: Patient Centered Outcomes Research Institute)
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Results first posted 2016-08-26 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-05

CONDITIONS: HPV Vaccination Status
Keywords: HPV vaccination; Tailored health messaging

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tailored intervention (Experimental): Intervention: tailored educational materials. In this arm, participants will complete a baseline survey on an iPad, view a series of educational webpages on the iPad, and complete a brief post intervention survey.
  Interventions: Behavioral: Tailored educational materials
- Untailored Intervention (Other): Intervention: untailored educational materials. In this arm, patients will view educational information on the iPad that is not responsive to their baseline questionnaire answers.
  Interventions: Behavioral: Untailored educational materials
- Usual Care (Other): Intervention: survey-only. Participants in the usual care arm will not view any educational materials or complete the baseline survey.
  Interventions: Behavioral: Survey-only

INTERVENTIONS:
Behavioral: Tailored educational materials — The tailored intervention will use participants' baseline survey responses to generate tailored educational messages about the HPV vaccine. These educational messages will reflect the top concerns indicated by the participant about the HPV vaccine. Additional tailoring will occur in the form of images matched to self-reported race and age, and using participants' first name in the information presented.
  Arms: Tailored intervention
Behavioral: Untailored educational materials — The untailored intervention will present educational information on the iPad that is not responsive to participants' baseline questionnaire answers and instead is derived directly from the HPV "Vaccine Information Sheet" that has been created by the Centers for Disease Control and Prevention.
  Arms: Untailored Intervention
Behavioral: Survey-only — Those in the usual care arm will be provided with a paper version of the Post Intervention Survey. This will be provided to participants after their clinic visit is completed.
  Arms: Usual Care

SUMMARY:
The purpose of this study is to evaluate an innovative approach to improving HPV vaccination among the Hispanic population. The clinical objectives/aims of this HPV educational intervention project are to determine:

1. The number of young adults and adolescents in each arm who received any dose of the HPV vaccine during the study period,
2. The number of young adults and adolescents in each arm who initiated the HPV vaccine series during the study period,
3. The number of young adults and adolescents in each arm who initiated but did not complete the HPV vaccine series during the study period,
4. The number of young adults and adolescents in each arm, among all eligible, who completed the HPV vaccine series during the study period,
5. The number of young adults and adolescents in each arm who completed the HPV vaccine series during the study period, among those who initiated the series at study start, and
6. The number of young adults and adolescents in each arm who completed the HPV vaccine series among those who initiated the series during the study period.

The implementation of this educational intervention in clinic waiting rooms is intended to assist primary care providers in communicating HPV vaccine awareness and education to parents and patients in a culturally tailored format.

DETAILED DESCRIPTION:
While HPV infection is nearly ubiquitous among the sexually active population, the morbidity and mortality from HPV-related diseases disproportionately affects minorities and the poor. Hispanic women are at particularly high risk as they have the highest rates of invasive cervical cancer when compared to all other racial or ethnic groups in the U.S. Initiating the 3-dose HPV vaccination series is more common among Hispanic adolescents than whites, but series completion has been lowest among Hispanic populations.

To understand barriers to HPV vaccination and to provide insight into ways in which an existing educational intervention should be modified for a Hispanic population, the investigators conducted focus groups among Hispanic parents and Latina young adults. All groups reported vaccine cost, access to insurance, and a general lack of awareness and/or understanding of either HPV or the vaccine as barriers. All groups also wanted substantially more "general" information about both HPV and the vaccine in order to make informed vaccination decisions. The educational intervention was generally well received but there were universal suggestions from all the groups to provide additional basic information about HPV infection, to add information about the vaccine for boys/young men, and to modify the color scheme and logo to make it more eye-catching and pleasing.

This current phase of the project will be comprised of real world testing of an iPad-based educational intervention about HPV, "Combatting HPV Infection and Cancer" (CHICOS) that has been revised and developed per focus group feedback to target the Hispanic population.

By providing information that patients and parents have clearly indicated they want in a way that is culturally sensitive and meaningful and also individually personalized, the investigators hope to improve HPV vaccination rates.

ELIGIBILITY:
Inclusion Criteria:

1. Parents of an adolescent between the ages of 9-17; OR a young adult patient between the ages of 18-26;
2. Adolescent/young adult has not yet received all three doses of the HPV vaccine.
3. Parent/young adult can read and converse in either English or Spanish

Exclusion Criteria:

1. Age <18,
2. Prisoners
3. Decisionally challenged subjects
4. Those who cannot read and converse in either English or Spanish
5. Those who have received all 3 doses of the HPV vaccine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1294 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda F Dempsey, MD, PhD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

REFERENCES:
- [Derived] Dempsey AF, Maertens J, Sevick C, Jimenez-Zambrano A, Juarez-Colunga E. A randomized, controlled, pragmatic trial of an iPad-based, tailored messaging intervention to increase human papillomavirus vaccination among Latinos. Hum Vaccin Immunother. 2019;15(7-8):1577-1584. doi: 10.1080/21645515.2018.1559685. Epub 2019 Feb 20. PMID 30689494

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Parent and young adult participants were recruited between June of 2014 and September of 2015 from one of five family health care clinics.
  Enrollment for the study was facilitated by 1) self-referral (passive recruitment), and 2) approach by research assistants (active recruitment).
Pre-assignment Details: Eligibility:
  1. Parents of an adolescent between the ages of 9-17; OR a young adult patient between the ages of 18-26;
  2. Adolescent/young adult has not yet received all three doses of the HPV vaccine;
  3. Parent/young adult can read and converse in either English or Spanish
Period: Overall Study
Arm/Group | Tailored Intervention | Untailored Intervention | Usual Care
Started | 430 | 425 | 439
Completed | 370 | 373 | 398
Not Completed | 60 | 52 | 41
Not completed — No match to vaccination records | 60 | 52 | 41

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tailored Intervention | Untailored Intervention | Usual Care | Total
Number analyzed (Participants) | 430 | 425 | 439 | 1294
Age, Continuous [Median (Full Range); unit: Years] — Population: Row population differs from overall, because young adult and adolescent groups were analyzed separately.
  Years
    Young Adults: number analyzed (Participants) | 143 | 151 | 152 | 446
    Young Adults | 22 [18 to 26] | 23 [18 to 26] | 23 [18 to 26] | 22 [18 to 26]
    Adolescents: number analyzed (Participants) | 287 | 274 | 287 | 848
    Adolescents | 12 [9 to 17] | 12 [9 to 17] | 12 [9 to 17] | 12 [9 to 17]
Sex/Gender, Customized [Number; unit: participants] — Population: Row population differs from overall because young adults and adolescents were analyzed separately.
  participants
    Female Young Adults: number analyzed (Participants) | 143 | 151 | 152 | 446
    Female Young Adults | 143 | 151 | 152 | 446
    Male Young Adults | 0 | 0 | 0 | 0
    Female Adolescents: number analyzed (Participants) | 287 | 274 | 287 | 848
    Female Adolescents | 143 | 133 | 139 | 415
    Male Adolescents: number analyzed (Participants) | 287 | 274 | 287 | 848
    Male Adolescents | 144 | 141 | 148 | 433
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Number of people that indicated "yes" I consider myself Hispanic/Latino. Population: Row population differs from overall because young adults and adolescents were analyzed separately.
  Participants
    Self-Identify Hispanic Young Adults: number analyzed (Participants) | 143 | 151 | 152 | 446
    Self-Identify Hispanic Young Adults | 123 | 127 | 130 | 380
    Self-Identify Hispanic Adolescents: number analyzed (Participants) | 287 | 274 | 287 | 848
    Self-Identify Hispanic Adolescents | 266 | 254 | 269 | 789
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Row population differs from overall because young adults and adolescents were analyzed separately.
  Participants
    White Non-Hispanic Young Adults: number analyzed (Participants) | 143 | 151 | 152 | 446
    White Non-Hispanic Young Adults | 17 | 20 | 19 | 56
    Other Race Young Adults: number analyzed (Participants) | 143 | 151 | 152 | 446
    Other Race Young Adults | 3 | 4 | 3 | 10
    White Non-Hispanic Adolescents: number analyzed (Participants) | 287 | 274 | 287 | 848
    White Non-Hispanic Adolescents | 18 | 19 | 17 | 54
    Other Race Adolescents: number analyzed (Participants) | 287 | 274 | 287 | 848
    Other Race Adolescents | 3 | 1 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 430 | 425 | 439 | 1294

OUTCOME MEASURES:

1. Primary Outcome: Number of Young Adults Who Received Any Dose of the HPV Vaccine During the Study Period
Description: This outcome describes the number of young adult participants between the ages of 18-26 who received any dose of the HPV vaccine during the study period.
Time Frame: 16 months
Population: Includes young adults in the sample who could be matched to vaccination data and had not received all 3 doses of the HPV vaccine prior to baseline.
Measure: Number; unit: participants
Arm/Group | Tailored Intervention | Untailored Intervention | Usual Care
Number analyzed (Participants) | 143 | 151 | 152
participants | 8 | 9 | 3
Statistical Analysis 1: Comparison: Tailored Intervention vs Untailored Intervention vs Usual Care; Test type: Superiority or Other; p = .36, Fisher Exact
Statistical Analysis 2: Comparison: Untailored Intervention vs Usual Care; Test type: Superiority or Other; p = .18, Fisher Exact
Statistical Analysis 3: Comparison: Tailored Intervention vs Usual Care; Test type: Superiority or Other; p = .22, Fisher Exact
Statistical Analysis 4: Comparison: Tailored Intervention vs Untailored Intervention; Test type: Superiority or Other; p = .88, Fisher Exact

2. Primary Outcome: Number of Young Adults Who Initiated the HPV Vaccine Series During the Study Period
Description: This outcome describes the number of young adult participants between the ages of 18-26 who had 0 doses of the HPV vaccine at study enrollment and received at least one dose during the study period.
Time Frame: 16 months
Population: Includes young adults in the sample who could be matched to vaccination data, who had not received all 3 doses of the HPV vaccine prior to baseline, and who also had 0 doses of the HPV vaccine prior to baseline.
Measure: Number; unit: participants
Arm/Group | Tailored Intervention | Untailored Intervention | Usual Care
Number analyzed (Participants) | 87 | 110 | 106
participants | 7 | 4 | 3
Statistical Analysis 1: Comparison: Tailored Intervention vs Untailored Intervention vs Usual Care; Test type: Superiority or Other; p = 0.35, Fisher Exact
Statistical Analysis 2: Comparison: Untailored Intervention vs Usual Care; Test type: Superiority or Other; p = 1.0, Fisher Exact
Statistical Analysis 3: Comparison: Tailored Intervention vs Usual Care; Test type: Superiority or Other; p = .23, Fisher Exact
Statistical Analysis 4: Comparison: Tailored Intervention vs Untailored Intervention; Test type: Superiority or Other; p = .23, Fisher Exact

3. Primary Outcome: Number of Young Adults Who Initiated But Did Not Complete the HPV Vaccine Series During the Study Period
Description: This outcome describes the number of young adult participants between the ages of 18-26 who had 0 doses of the HPV vaccine at study enrollment and did not complete the vaccine series during the study period.
Time Frame: 16 months
Population: Includes young adults in the sample who could be matched to vaccination data, who had not received all 3 doses of the HPV vaccine prior to baseline, and who also had 0 doses of the HPV vaccine prior to baseline and did not complete the vaccine series during the study period.
Measure: Number; unit: participants
Arm/Group | Tailored Intervention | Untailored Intervention | Usual Care
Number analyzed (Participants) | 11 | 12 | 11
participants | 9 | 12 | 6
Statistical Analysis 1: Comparison: Tailored Intervention vs Untailored Intervention vs Usual Care; Test type: Superiority or Other; p = 0.37, Fisher Exact
Statistical Analysis 2: Comparison: Untailored Intervention vs Usual Care; Test type: Superiority or Other; p = .23, Fisher Exact
Statistical Analysis 3: Comparison: Tailored Intervention vs Usual Care; Test type: Superiority or Other; p = .25, Fisher Exact
Statistical Analysis 4: Comparison: Tailored Intervention vs Untailored Intervention; Test type: Superiority or Other; p = .70, Fisher Exact

4. Primary Outcome: Number of Young Adults, Among All Eligible, Who Completed the HPV Vaccine Series During the Study Period
Description: This outcome describes the number of young adult participants between the ages of 18-26 who had 0, 1 or 2 doses of the HPV vaccine at study enrollment and completed the vaccine series during the study period.
Time Frame: 16 months
Population: Includes young adults in the sample who could be matched to vaccination data, who had not received all 3 doses of the HPV vaccine prior to baseline, and who also had 0, 1 or 2 doses of the HPV vaccine at study enrollment and completed the vaccine series during the study period.
Measure: Number; unit: participants
Arm/Group | Tailored Intervention | Untailored Intervention | Usual Care
Number analyzed (Participants) | 100 | 120 | 117
participants | 1 | 4 | 2
Statistical Analysis 1: Comparison: Tailored Intervention vs Untailored Intervention vs Usual Care; Test type: Superiority or Other; p = 0.59, Fisher Exact
Statistical Analysis 2: Comparison: Untailored Intervention vs Usual Care; Test type: Superiority or Other; p = .52, Fisher Exact
Statistical Analysis 3: Comparison: Tailored Intervention vs Usual Care; Test type: Superiority or Other; p = .71, Fisher Exact
Statistical Analysis 4: Comparison: Tailored Intervention vs Untailored Intervention; Test type: Superiority or Other; p = .34, Fisher Exact

5. Primary Outcome: Number of Young Adults Who Completed the HPV Vaccine Series During the Study Period, Among Those Who Initiated the Series at Study Start
Description: This outcome describes the number of young adult participants between the ages of 18-26 who had 1 or 2 doses of the HPV vaccine at study enrollment and completed the vaccine series during the study period.
Time Frame: 16 months
Population: Includes young adults in the sample who could be matched to vaccination data, who had not received all 3 doses of the HPV vaccine prior to baseline, and who also had 1 or 2 doses of the HPV vaccine at study enrollment and completed the vaccine series during the study period.
Measure: Number; unit: participants
Arm/Group | Tailored Intervention | Untailored Intervention | Usual Care
Number analyzed (Participants) | 31 | 36 | 42
participants | 0 | 4 | 0
Statistical Analysis 1: Comparison: Tailored Intervention vs Untailored Intervention vs Usual Care; Test type: Superiority or Other; p = 0.16, Fisher Exact
Statistical Analysis 2: Comparison: Untailored Intervention vs Usual Care; Test type: Superiority or Other; p = .15, Fisher Exact
Statistical Analysis 3: Comparison: Tailored Intervention vs Usual Care; Test type: Superiority or Other; p = .98, Fisher Exact
Statistical Analysis 4: Comparison: Tailored Intervention vs Untailored Intervention; Test type: Superiority or Other; p = .34, Fisher Exact

6. Primary Outcome: Number of Young Adults Who Completed the HPV Vaccine Series Among Those Who Initiated the Series During the Study Period
Description: This outcome describes the number of young adult participants between the ages of 18-26 who had 0 doses of the HPV vaccine at study enrollment and completed the vaccine series during the study period.
Time Frame: 16 months
Population: Includes young adults in the sample who could be matched to vaccination data, who had not received all 3 doses of the HPV vaccine prior to baseline, and who also had 0 doses of the HPV vaccine at study enrollment and completed the vaccine series during the study period.
Measure: Number; unit: participants
Arm/Group | Tailored Intervention | Untailored Intervention | Usual Care
Number analyzed (Participants) | 11 | 12 | 11
participants | 2 | 0 | 5
Statistical Analysis 1: Comparison: Tailored Intervention vs Untailored Intervention vs Usual Care; Test type: Superiority or Other; p = 0.37, Fisher Exact
Statistical Analysis 2: Comparison: Untailored Intervention vs Usual Care; Test type: Superiority or Other; p = .23, Fisher Exact
Statistical Analysis 3: Comparison: Tailored Intervention vs Usual Care; Test type: Superiority or Other; p = .25, Fisher Exact
Statistical Analysis 4: Comparison: Tailored Intervention vs Untailored Intervention; Test type: Superiority or Other; p = .70, Fisher Exact

7. Primary Outcome: Number of Adolescents Who Received Any Dose of the HPV Vaccine During the Study Period
Description: This outcome describes the number of adolescent participants between the ages of 9-17 who received any dose of the HPV vaccine during the study period.
Time Frame: 16 months
Population: Includes adolescents in the sample who could be matched to vaccination data and had not received all 3 doses of the HPV vaccine prior to baseline.
Measure: Number; unit: participants
Arm/Group | Tailored Intervention | Untailored Intervention | Usual Care
Number analyzed (Participants) | 287 | 274 | 287
participants | 124 | 122 | 121
Statistical Analysis 1: Comparison: Tailored Intervention vs Untailored Intervention vs Usual Care; Test type: Superiority or Other; p = 0.87, Chi-squared
Statistical Analysis 2: Comparison: Untailored Intervention vs Usual Care; Test type: Superiority or Other; p = 0.62, Chi-squared
Statistical Analysis 3: Comparison: Tailored Intervention vs Usual Care; Test type: Superiority or Other; p = 0.81, Chi-squared
Statistical Analysis 4: Comparison: Tailored Intervention vs Untailored Intervention; Test type: Superiority or Other; p = 0.76, Chi-squared

8. Primary Outcome: Number of Adolescents Who Initiated the HPV Vaccine Series During the Study Period
Description: This outcome describes the number of adolescent participants between the ages of 9-17 who had 0 doses of the HPV vaccine at study enrollment and received at least one dose during the study period.
Time Frame: 16 months
Population: Includes adolescents in the sample who could be matched to vaccination data, who had not received all 3 doses of the HPV vaccine prior to baseline, and who also had 0 doses of the HPV vaccine prior to baseline.
Measure: Number; unit: participants
Arm/Group | Tailored Intervention | Untailored Intervention | Usual Care
Number analyzed (Participants) | 187 | 174 | 197
participants | 74 | 73 | 75
Statistical Analysis 1: Comparison: Tailored Intervention vs Untailored Intervention vs Usual Care; Test type: Superiority or Other; p = 0.70, Chi-squared
Statistical Analysis 2: Comparison: Untailored Intervention vs Usual Care; Test type: Superiority or Other; p = 0.41, Chi-squared
Statistical Analysis 3: Comparison: Tailored Intervention vs Usual Care; Test type: Superiority or Other; p = 0.59, Chi-squared
Statistical Analysis 4: Comparison: Tailored Intervention vs Untailored Intervention; Test type: Superiority or Other; p = 0.74, Chi-squared

9. Primary Outcome: Number of Adolescents Who Initiated But Did Not Complete the HPV Vaccine Series During the Study Period
Description: This outcome describes the number of adolescent participants between the ages of 9-17 who had 0 doses of the HPV vaccine at study enrollment and did not complete the vaccine series during the study period.
Time Frame: 16 months
Population: Includes adolescents in the sample who could be matched to vaccination data, who had not received all 3 doses of the HPV vaccine prior to baseline, and who also had 0 doses of the HPV vaccine prior to baseline and did not complete the vaccine series during the study period.
Measure: Number; unit: participants
Arm/Group | Tailored Intervention | Untailored Intervention | Usual Care
Number analyzed (Participants) | 103 | 106 | 125
participants | 79 | 93 | 89
Statistical Analysis 1: Comparison: Tailored Intervention vs Untailored Intervention vs Usual Care; Test type: Superiority or Other; p = 0.38, Chi-squared
Statistical Analysis 2: Comparison: Untailored Intervention vs Usual Care; Test type: Superiority or Other; p = 0.17, Chi-squared
Statistical Analysis 3: Comparison: Tailored Intervention vs Usual Care; Test type: Superiority or Other; p = 0.60, Chi-squared
Statistical Analysis 4: Comparison: Tailored Intervention vs Untailored Intervention; Test type: Superiority or Other; p = 0.35, Chi-squared

10. Primary Outcome: Number of Adolescents, Among All Eligible, Who Completed the HPV Vaccine Series During the Study Period
Description: This outcome describes the number of adolescent participants between the ages of 9-17 who had 0, 1 or 2 doses of the HPV vaccine at study enrollment and completed the vaccine series during the study period.
Time Frame: 16 months
Population: Includes adolescents in the sample who could be matched to vaccination data, who had not received all 3 doses of the HPV vaccine prior to baseline, and who also had 0, 1 or 2 doses of the HPV vaccine at study enrollment and completed the vaccine series during the study period.
Measure: Number; unit: participants
Arm/Group | Tailored Intervention | Untailored Intervention | Usual Care
Number analyzed (Participants) | 233 | 229 | 241
participants | 54 | 39 | 48
Statistical Analysis 1: Comparison: Tailored Intervention vs Untailored Intervention vs Usual Care; Test type: Superiority or Other; p = 0.39, Chi-squared
Statistical Analysis 2: Comparison: Untailored Intervention vs Usual Care; Test type: Superiority or Other; p = 0.51, Chi-squared
Statistical Analysis 3: Comparison: Tailored Intervention vs Usual Care; Test type: Superiority or Other; p = 0.49, Chi-squared
Statistical Analysis 4: Comparison: Tailored Intervention vs Untailored Intervention; Test type: Superiority or Other; p = 0.14, Chi-squared

11. Primary Outcome: Number of Adolescents Who Completed the HPV Vaccine Series During the Study Period, Among Those Who Initiated the Series at Study Start
Description: This outcome describes the number of adolescent participants between the ages of 9-17 who had 1 or 2 doses of the HPV vaccine at study enrollment and completed the vaccine series during the study period.
Time Frame: 16 months
Population: Includes adolescents in the sample who could be matched to vaccination data, who had not received all 3 doses of the HPV vaccine prior to baseline, and who also had 1 or 2 doses of the HPV vaccine at study enrollment and completed the vaccine series during the study period.
Measure: Number; unit: participants
Arm/Group | Tailored Intervention | Untailored Intervention | Usual Care
Number analyzed (Participants) | 140 | 145 | 165
participants | 59 | 41 | 55
Statistical Analysis 1: Comparison: Tailored Intervention vs Untailored Intervention vs Usual Care; Test type: Superiority or Other; p = 0.09, Chi-squared
Statistical Analysis 2: Comparison: Untailored Intervention vs Usual Care; Test type: Superiority or Other; p = 0.51, Chi-squared
Statistical Analysis 3: Comparison: Tailored Intervention vs Usual Care; Test type: Superiority or Other; p = 0.15, Chi-squared
Statistical Analysis 4: Comparison: Tailored Intervention vs Untailored Intervention; Test type: Superiority or Other; p = 0.03, Chi-squared

12. Primary Outcome: Number of Adolescents Who Completed the HPV Vaccine Series Among Those Who Initiated the Series During the Study Period
Description: This outcome describes the number of adolescent participants between the ages of 9-17 who had 0 doses of the HPV vaccine at study enrollment and completed the vaccine series during the study period.
Time Frame: 16 months
Population: Includes adolescents in the sample who could be matched to vaccination data, who had not received all 3 doses of the HPV vaccine prior to baseline, and who also had 0 doses of the HPV vaccine at study enrollment and completed the vaccine series during the study period.
Measure: Number; unit: participants
Arm/Group | Tailored Intervention | Untailored Intervention | Usual Care
Number analyzed (Participants) | 103 | 106 | 125
participants | 24 | 13 | 36
Statistical Analysis 1: Comparison: Tailored Intervention vs Untailored Intervention vs Usual Care; Test type: Superiority or Other; p = 0.38, Chi-squared
Statistical Analysis 2: Comparison: Untailored Intervention vs Usual Care; Test type: Superiority or Other; p = 0.17, Chi-squared
Statistical Analysis 3: Comparison: Tailored Intervention vs Usual Care; Test type: Superiority or Other; p = 0.60, Chi-squared
Statistical Analysis 4: Comparison: Tailored Intervention vs Untailored Intervention; Test type: Superiority or Other; p = 0.35, Chi-squared

ADVERSE EVENTS:
Time Frame: 16 months
Groups:
- Usual Care: Intervention: Survey-only. Intervention: survey-only. Participants in the usual care arm will not view any educational materials or complete the baseline survey.
  Survey-only: Those in the usual care arm will be provided with a paper version of the Post Intervention Survey. This will be provided to participants after their clinic visit is completed.
Arm/Group | Tailored Intervention | Untailored Intervention | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/430 | 0/425 | 0/439
Other Adverse Events (participants affected / at risk) | 0/430 | 0/425 | 0/439

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes